CLINICAL TRIAL: NCT00311935
Title: Randomized Controlled Trial of Laparoscopic vs. Open Mesh Inguinal Hernia Repair in Men Under the Age of 60
Brief Title: Laparoscopic vs Open Hernia Mesh Repair for Inguinal Hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Waitemata District Health Board (Other Government)
Collaborators: Tyco Healthcare Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hernia repair study
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Hernia, Inguinal
Keywords: Hernia; Inguinal; Groin; Laparoscopic; Open; Abdominal wall
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: method of hernia repair

SUMMARY:
This study will determine whether laparoscopic and open hernia repair have the same recurrence and complication rates in the under 60yr old age group. The overall financial costs of each repair will also be compared.

DETAILED DESCRIPTION:
Study population is Waitemata Health (Auckland New Zealand) patients presenting to clinic with unilateral primary inguinal hernia aged less than 60 years, fit for surgery and able to consent for the study. Randomized to open mesh repair or laparoscopic preperitoneal mesh repair. Two surgeons (Dr Rodgers and Dr Hammodat) using a standardized technique. Conversion rates from lap to open will be recorded.

Phone assessment postop day 1, 1 week and at 6 months. Clinic assessment at 4 weeks, 1 year and 2 years.

Primary outcome is hernia recurrence which will be assessed by a research nurse independent of surgeon at each clinic appointment. Assessment to also include assessment of ongoing symptoms such as pain/discomfort, sensory disturbance, and sexual dysfunction.

Quality of life assessment (SF 36 questionnaire) preoperatively and at each assessment.

Pain assessment 4hrs postop and at all other assessments by score 0-10 and measurement of pain relief.

Cost analysis to include the following parameters: theatre equipment costs, theatre time, drug use, hospital stay, time to return to work, time to return to normal activities.

Interim analysis at 2 years of followup by independent Health and Safety committee. Final analysis at 4 years of followup.

ELIGIBILITY:
Inclusion Criteria:

* Male <60yrs with primary inguinal hernia

Exclusion Criteria:

* Recurrent hernia
* Bilateral hernia
* Non-reducible/obstructed hernia
* Previous lower abdominal surgery/radiotherapy

Ages: 15 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Estimated)
Dates: Start 2006-04; Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence rates at 2 years post surgery.

SECONDARY OUTCOMES:
Complication rates.
Duration of procedure.
Cost of equipment use.
Rate of conversion to open procedure
Length of hospital stay.
Time to return to work and usual activities.
Pain scores and analgesic use.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rodgers, MBCHB,FRACS, Principal Investigator — Waitemata District Health Board
Locations (1):
- Waitemata District Health Board, Auckland, New Zealand